CLINICAL TRIAL: NCT01338597
Title: Clinical Benefits of Reduced Subcutaneous Dissection in Endoscopic Thyroidectomy
Brief Title: Impact of Dissection Area on the Clinical Outcome of Endoscopic Thyroidectomy
Acronym: ET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Military Medical University (Other)
Responsible Party: department of general surgery, changzheng hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMMU-2011-ET-1
Record Dates: First submitted 2011-04-11; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Thyroid Tumor
Keywords: thyroidectomy; invasiveness
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard (Experimental): 3 trocars are needed. two in the circumareolar region and one in the parasternal region. the dissection area begins from the trocar site and extends to the neck.
  Interventions: Procedure: endoscopic thyroidectomy
- limited dissection (Experimental): the dissection is reduced by creating a long tunnel from the trocar site and the dissection area confined in the upper chest wall and in the neck.
  Interventions: Procedure: endoscopic thyroidectomy

INTERVENTIONS:
Procedure: endoscopic thyroidectomy — endoscopic thyroidectomy via the breast approach. the difference between two arms is in the subcutaneous dissection area.
  Other Names: limited flap dissection endoscopic thyroidectomy

SUMMARY:
The purpose of this study is to investigate whether reduced subcutaneous dissection area could offer patients more clinical benefits.

DETAILED DESCRIPTION:
To create a working place in the chest wall is an inevitable step of endoscopic thyroidectomy. Large subcutaneous area was considered a drawback of endoscopic thyroidectomy. The purpose of this study is to investigate whether subcutaneous dissection area has influence on clinical outcome of endoscopic thyroidectomy, such as post-operative pain, complication rate and post-operative discomfort.

ELIGIBILITY:
Inclusion Criteria:

* thyroid nodule diagnosed by ultrasound
* willing to undergo endoscopic thyroidectomy

Exclusion Criteria:

* conversion to open surgery
* unwilling to join the research

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
post-operative pain | 24h post-operation
  24hs after operation, post-operative pain is evaluated by VAS(visual analoge scale)

SECONDARY OUTCOMES:
number of patients with adverse effect | within 3 months after surgery
  record how many patients had adverse effects(eg. bruise, seroma, hematoma, hoarseness,hypocalciemia)

CONTACTS AND LOCATIONS:
Overall Officials: ming qiu, MD, Study Chair — Changzheng Hospital
Locations (1):
- Department of General Surgery, Changzheng Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Wang M, Zhang T, Mao Z, Dong F, Li J, Lu A, Hu W, Zang L, Jiang Y, Zheng M. Effect of endoscopic thyroidectomy via anterior chest wall approach on treatment of benign thyroid tumors. J Laparoendosc Adv Surg Tech A. 2009 Apr;19(2):149-52. doi: 10.1089/lap.2008.0296. PMID 19361288